CLINICAL TRIAL: NCT03099031
Title: Prediction of Thromboembolic Recurrences in Cancer Patients With Venous Thromboembolic Disease (TED)
Brief Title: Non Interventional Study of the Validation of the Ottawa Score in Cancer Patients With Venous Thromboembolism (VTE)
Acronym: PREDICARE
Status: Completed | Type: Observational
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-INNOHEP-1093
Record Dates: First submitted 2017-03-01; First posted 2017-04-04 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Venous Thromboembolism
Keywords: Ottawa score; tinzaparin; low-molecular weight heparin; anticoagulants; venous thrombosis; thromboembolism; hemostatic disorders; vascular disease; neoplasms; breast neoplasms; lung neoplasms; prostatic neoplasms; colorectal neoplasms; genital neoplasms; urogenital neoplasms; intestinal neoplasms; digestive system neoplasms; lymphoma; leukemia; multiple myeloma; lymphoproliferative disorders; myeloproliferative disorders; lymphatic disease
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Thromboembolism; Hemostatic Disorders; Vascular Diseases; Neoplasms; Breast Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms; Urogenital Neoplasms; Intestinal Neoplasms; Digestive System Neoplasms; Lymphoma; Leukemia; Multiple Myeloma; Lymphoproliferative Disorders; Myeloproliferative Disorders; Lymphatic Diseases | interventions — Tinzaparin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tinzaparin: Patients with objectively confirmed cancer associated venous thromboembolism receiving tinzaparin treatment to prevent recurrence of venous thromboembolism
  Interventions: Drug: Tinzaparin

INTERVENTIONS:
Drug: Tinzaparin — Subcutaneous injection of 175 IU/kg once daily for 6 months
  Other Names: Innohep®

SUMMARY:
The purpose of this study is to validate the Ottawa score (risk of thromboembolic recurrences) in cancer patients with thromboembolic disease treated with tinzaparin (Innohep®)

DETAILED DESCRIPTION:
The Ottawa score is a clinical predictive score aiming at stratifying thromboembolic recurrences in cancer patients according to identified clinical risk factors and histological type of the tumor. This score has never been validated externally in a prospective way in patients treated with tinzaparin. The objective of this observational prospective study is to enroll cancer patients with TED treated with tinzaparin for a planned period of 6 months and to collect data on thromboembolic recurrences, major hemorrhages, deaths and heparin-induced thrombocytopenia

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients with histologically confirmed, active or evolving, solid or liquid tumour, or
* Suspected malignant tumour confirmed within a month of index VTE occurrence
* Treated with specific metastatic or adjuvant anti-cancer treatment
* Patients with recent diagnosis of documented symptomatic or incidental VTE and a prescription of tinzaparin for 6 months
* Proximal or distal VTE of lower limbs
* Pulmonary embolism
* Inferior or superior vena cava thrombosis
* Iliac vein thrombosis

Exclusion Criteria:

* Skin cancer other than melanoma
* Life expectancy less than 6 months
* Superficial isolated thrombosis
* Isolated subsegmental pulmonary embolism
* Cerebral, visceral thrombosis
* Superior limbs VTE or Central catheter thrombosis
* Patients being treated with anticoagulants by more than 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient population from French general hospitals, anticancer centres, and university hospitals treating more than 1000 cancer patients per year
Sampling Method: Probability Sample
Enrollment: 420 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-05-15 (Actual)

PRIMARY OUTCOMES:
Venous thromboembolism recurrence | 6 months

SECONDARY OUTCOMES:
Major hemorrhage | 6 months
Death | 6 months
  All cause mortality
Heparin induced thrombocytopenia | 6 months

OTHER OUTCOMES:
Premature treatment discontinuation | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: G Meyer, Professor, Principal Investigator — Service de pneumologie et de soins intensifs, Hôpital Européen Georges Pompidou, Paris; F Scotte, Dr, Principal Investigator — Unité fonctionnelle de soins oncologiques de support, Hôpital Européen Georges Pompidou, Paris
Locations (1):
- George Pompidou European Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No